CLINICAL TRIAL: NCT01014884
Title: Coventry Outcomes Study of Seniors: A Dual-arm, Controlled, Randomized, Comparative Effectiveness Study to Evaluate the Effect of a Multidisciplinary Team's Intervention Versus Usual Care on the Incidence of Nonelective Hospitalizations in a Medicare Population
Brief Title: Coventry Outcomes Study of Seniors (COSS): A Comparative Effectiveness Study to Evaluate the Effect of a Multidisciplinary Team's Intervention on the Incidence of Nonelective Hospitalizations in a Medicare Population
Acronym: COSS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated by Sponsor
Sponsor: Medco Health Solutions, Inc. (Industry)
Collaborators: Coventry Health Care, Inc. (Industry)
Responsible Party: Julia O. McEacherm, Research Director, Medco Health Solutions, Inc.
Other Study IDs: 7714
Record Dates: First submitted 2009-11-12; First posted 2009-11-17 (Estimated); Last update posted 2010-01-21 (Estimated); Status verified 2010-01

CONDITIONS: Heart Failure; Chronic Obstructive Pulmonary Disease; Cardiovascular Disease; Diabetes; Osteoporosis
MeSH Terms: conditions — Heart Failure; Pulmonary Disease, Chronic Obstructive; Cardiovascular Diseases; Diabetes Mellitus; Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Other): The control group will receive usual care as provided by your Health Plan.
  Interventions: Other: Usual case management and pharmacy management as provided by the health Plan and the pharmacy benefit manager
- Intervention group (Other): Additional visits will be conducted by a member of the multidisciplinary team (case manager/nurse, social worker and/or pharmacist that will be either face to face or by telephone.
  Interventions: Other: Multidisciplinary team interventions; Other: Multidisciplinary team bimonthly visits either in person or via telephone.

INTERVENTIONS:
Other: Multidisciplinary team interventions — The multidisciplinary team will determine which intervention should be applied to the participant in the intervention group based on their health risk assessment responses as well as medication review and visual inspection of the home.
  Arms: Intervention group
Other: Multidisciplinary team bimonthly visits either in person or via telephone.
  Arms: Intervention group
Other: Usual case management and pharmacy management as provided by the health Plan and the pharmacy benefit manager
  Arms: Control Group

SUMMARY:
The investigators are studying the impact of the interventions of a multidisciplinary team (MDT) - consisting of a Coventry case manager, social worker, and medical director, alongside a Medco specialist pharmacist - on the hospitalization rates of high risk seniors with chronic conditions, compared with a usual care approach. The study will also examine the impact on quality of life, medication adherence, medical costs, hospital readmission rates, and a variety of other important measures. The outcome of COSS may support a means to further enhance and develop a comprehensive care model program by leveraging the partnership between a health plan and a pharmacy benefit manager.

DETAILED DESCRIPTION:
The multidisciplinary team will provide face-to-face visits in a home setting with interventions that focus on five key areas: care transitions, self-management, care coordination, pharmacy and prevention, all designed to support high-risk Medicare members and their relationship with their primary care providers. If the study proves to reduce hospitalizations in the senior population, it could provide important guidance for future efforts to reduce the cost and improve the quality of care for seniors with chronic conditions.

ELIGIBILITY:
Inclusion Criteria:

* Inouye Risk Score >3 calculated on Coventry Claims
* Medicare Advantage beneficiaries age > 65 years
* Continuous eligibility > 12 months prior to study
* Ability to be contacted via telephone
* Subject is willing and able to provide informed consent
* Willing to comply with all study procedures and be available for the duration of the study

Exclusion Criteria:

* Active cancer treatment (i.e. chemotherapy or radiation) in the past 6 months
* Living anywhere other than a community setting [i.e. Skilled nursing facility (SNF)]
* Just-In-Time (JIT) Members
* Members with a geographic location > 60 from either St. Louis or Kansas City, MO.
* Solid organ transplant recipients
* Active enrollment in another clinical research study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2150 (Estimated)
Dates: Start 2009-11; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Determine the impact of multidisciplinary team interventions in reducing the rate of non-elective hospitalizations over a 12 month period compared to usual care | 12 months

SECONDARY OUTCOMES:
Determine the impact of multidisciplinary team interventions on the rate of emergency room visits not resulting in hospitalization in a 24 hour period or less. | 12 months
Determine the impact of multidisciplinary team interventions versus usual care on health-related quality of life (HR-QOL) | 12 months
Determine the impact of MDT interventions versus usual care on inpatient costs associated with non-elective hospital events [rehabilitation, physician, incurred but not reported (IBNR)] | 12 months
Determine the impact of multidisciplinary team interventions versus usual care on total outpatient costs (physician, pharmacy,rehabilitation) | 12 months
Determine the impact of multidisciplinary team interventions versus usual care on satisfaction with care | 12 months
Determine the impact of multidisciplinary team interventions versus usual care on rate of non-elective hospitalizations by chronic condition | 12 months
Determine the impact of multidisciplinary team interventions versus usual care on non-elective hospital readmissions at 30, 60, and 90 days following the first non-elective hospitalization event | 12
Determine the impact of multidisciplinary team interventions versus usual care on the length of stay (LOS) of each non-elective hospitalization | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Julia O McEachern, MHS, PA-C, Principal Investigator — Medco Health Solutions, Inc.; Stephen L Cavalieri, MD, Principal Investigator — Coventry Health Care, Inc.
Locations (2):
- United States (2):
  - Kansas City, Missouri
  - St Louis, Missouri